CLINICAL TRIAL: NCT05900440
Title: Use of Artificial Intelligence for Acquisition of Limited Echocardiograms
Brief Title: Artificial Intelligence for Learning Point-of-Care Ultrasound
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andre Kumar, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-42094
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Education, Medical; Ultrasound Imaging
Keywords: Medical Education; Point-of-Care Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence Group (Experimental)
  Interventions: Other: Ultrasound with Artificial Inteligence Engabled
- Non Artificial Intelligence Group (Active Comparator)
  Interventions: Other: Ultrasound without Artificial Intelligence Enabled

INTERVENTIONS:
Other: Ultrasound with Artificial Inteligence Engabled — Participants shall be randomized 1:1 to receive personal access to a handheld ultrasound device with artificial intelligence vs a device with no artificial intelligence. The groups shall not cross over in which intervention they received.
  Arms: Artificial Intelligence Group
Other: Ultrasound without Artificial Intelligence Enabled — Participants shall be randomized 1:1 to receive personal access to a handheld ultrasound device with artificial intelligence vs a device with no artificial intelligence. The groups shall not cross over in which intervention they received.
  Arms: Non Artificial Intelligence Group

SUMMARY:
Point-of care-ultrasonography has the potential to transform healthcare delivery through its diagnostic and therapeutic utility. Its use has become more widespread across a variety of clinical settings as more investigations have demonstrated its impact on patient care. This includes the use of point-of-care ultrasound by trainees, who are now utilizing this technology as part of their diagnostic assessments of patients. However, there are few studies that examine how efficiently trainees can learn point-of-care ultrasound and which training methods are more effective. The primary objective of this study is to assess whether artificial intelligence systems improve internal medicine interns' knowledge and image interpretation skills with point-of-care ultrasound. Participants shall be randomized to receive personal access to handheld ultrasound devices to be used for learning with artificial intelligence vs devices with no artificial intelligence. The primary outcome will assess their interpretive ability with ultrasound images/videos. Secondary outcomes will include rates of device usage and performance on quizzes.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residents rotating on the general inpatient wards service.

Exclusion Criteria:

* Residents who had taken an ultrasound elective offered by our residency program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to acquire cardiac ultrasound images | During procedure (300 seconds)
  This will be measured as the time to acquire a cardiac ultrasound image on a standardized patient, measured in seconds.

SECONDARY OUTCOMES:
Assessment of the quality of captured images | During procedure (300 seconds)
  Participants will acquire cardiac ultrasound images on a standardized patient. Two reviewers will review the images and provide a numerical assessment of image quality based on the Rapid Assessment for Competency in Echocardiography (RACE) Scale. This is a 0-20 point scale, with higher scores denoting higher image quality (e.g. a better quality image).

CONTACTS AND LOCATIONS:
Overall Officials: Andre D Kumar, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Weng Y, Wang L, Bentley J, Almli M, Hom J, Witteles R, Ahuja N, Kugler J. Portable Ultrasound Device Usage and Learning Outcomes Among Internal Medicine Trainees: A Parallel-Group Randomized Trial. J Hosp Med. 2020 Feb 11;15(2):e1-e6. doi: 10.12788/jhm.3351. Online ahead of print. PMID 32118565